CLINICAL TRIAL: NCT01916525
Title: Effectiveness of Exercise-based Rehabilitation Program for Patients After Acute Coronary Syndrome
Brief Title: Effectiveness of Exercise Cardiac Rehabilitation
Acronym: EFEX-CARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Collaborators: Verve Research, Oulu, Finland (Other); University of Eastern Finland (Other); Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Mikko Tulppo, Adjunct professor, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Verve-139226
Record Dates: First submitted 2013-07-30; First posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Cost-effectiveness of Exercise-based Rehabilitation Program
Keywords: Acute coronary syndrome; Cost-effectiveness; Cardiac rehabilitation; Exercise; Physical activity; Home monitoring
MeSH Terms: conditions — Acute Coronary Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise based cardiac rehabilitation (Experimental): Patients will receive written instructions and a referral to the exercise-based rehabilitation unit. The patient will be taught to use fitness room. Each session of training will be controlled by heart rate. Instruction will also be given for at-home training and filling in a training diary, and training will be scheduled at Verve once a week. On the first visit the patient will receive a device that measures physical activity during the study. Training will also be monitored from the training diary. Structured questionnaires will be used to check compliance and implementation of care will be determined from medication and other health-related habits once a month (during the first 6 months) and finally after 12 months.
  Interventions: Behavioral: Exercise based cardiac rehabilitation
- Control (No Intervention): A conventional post-acute care group treated according to finnish guidelines.

INTERVENTIONS:
Behavioral: Exercise based cardiac rehabilitation — The cost-effectiveness between the exercise training vs. control groups
  Arms: Exercise based cardiac rehabilitation

SUMMARY:
The objective of this multidisciplinary study is to employ health-economic evaluation in determining the health benefits achieved with exercise-based cardiac rehabilitation and the costs derived from it compared with conventional post-acute care of cardiac patients in the Finnish health care system.

DETAILED DESCRIPTION:
The cost-effectiveness of exercise-based cardiac rehabilitation has not been systematically studied earlier in Finland, and it is not justifiable to directly apply the results of studies done in other countries to circumstances in Finland due to differences in the health care and social security systems between the countries. The research will utilize top Finnish expertise spanning clinical cardiology, health economics, and physical education. The hypothesis is that a quality-adjusted life year of a cardiac patient (cost/QALY) is 20 % less costly in a rehabilitation group than in a conventional post-acute care group.

The participants in the study will be recruited from Oulu University Hospital patients from the Oulu region (n = 300) who have suffered acute coronary syndrome (angiographically diagnosed coronary artery disease). Of these patients, 130 will be randomized to exercise-based cardiac rehabilitation (Verve) and 170 to a control group. Dropping out of the intervention will be mini-mized by means of careful definition of the inclusion criteria and close follow-up. The rehabilitation will seek to implement the most recent international recommendations for health-enhancing physical activity (% of those who achieved the exercise target). Instructions for a progressive training model will be compiled. The amount of exercise will be monitored objectively with a wrist-worn device based on wellness technology. Subjective loading of both the training and health-enhancing physical activity will be monitored using self-evaluation. The study will last one year for each patient, after which cost-effectiveness will be analyzed (University of Eastern Finland). The results of the research will facilitate decision making and choices in Finnish health care when arranging rehabilitation for cardiac patients and planning the optimal utilization of health care resources.

ELIGIBILITY:
Inclusion Criteria:

* The patients undergo coronary angiography and are diagnosed with coronary artery disease.

Exclusion Criteria:

* New York Heart Association (NYHA) class IV
* heart failure
* unstable chest pain (angina pectoris) at the time of randomization
* severe peripheral atherosclerosis (intermittent claudication)
* severe retinopathy or neuropathy related to diabetes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Cost / quality-adjusted life year of a cardiac patient (QALY) | One year / patient

SECONDARY OUTCOMES:
Major Adverse Cardiac Event (MACE) | One year / patient
  significant clinical adverse events, overall mortality, and acute cardiac arrest or resuscitation from cardiac arrest.

CONTACTS AND LOCATIONS:
Overall Officials: Mikko P Tulppo, PhD, Study Director — University of Oulu
Locations (1):
- Verve, Oulu, Finland